CLINICAL TRIAL: NCT06056245
Title: Postoperative Pharmacokinetics of Methadone in Patients With Chronic Kidney Disease
Brief Title: Methadone Pharmacokinetics in End-stage Renal Disease
Acronym: MCKD
Status: Recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 230125010
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Diseases; Post Operative Pain; Pain, Acute
Keywords: Methadone; Patient Controlled Anesthesia; Chronic Kidney Diseases; Post Operative Pain
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pain, Postoperative; Acute Pain | interventions — Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with chronic kidney disease (CKD) over 18 years old undergoing surgery using general anesthesia with subsequent use of intravenous patient-controlled analgesia (IV-PCA) of methadone.
  Interventions: Procedure: Preoperative step; Drug: Intraoperative; Drug: Post-operative

INTERVENTIONS:
Procedure: Preoperative step — * Explanation of the surgery and use of the IV-PCA pump.
  * Signed informed consent.
Drug: Intraoperative — Bolus of methadone 0.1mg/kg based on ideal body weight (up to a maximum dose of 20 mg), at the beginning of surgery.
  Other Names: Methadone administration during surgery
Drug: Post-operative — Installation of IV-PCA of methadone. Program to be used with no background infusion, boluses of 1 mg, and the intervals between boluses of 8 minutes.
  Other Names: Methadone boluses administered by IV-PCA pump

SUMMARY:
The goal of this observational study is to describe the influence of renal function on the pharmacokinetics of methadone used through an intravenous patient-controlled analgesia (IV-PCA) pump for the management of acute postoperative pain. After surgery the participants will use an IV-PCA of methadone and blood samples will be withdrawn to measure the plasmatic levels of it.

The main question the study aims to answer is:

• Is the pharmacokinetic of methadone used in an IV-PCA pump impaired in patients with chronic kidney disease?

DETAILED DESCRIPTION:
This study will be carried out at the Pontifical Catholic University of Chile Hospital with prior approval by the ethics committee. Study staff will assess the inclusion criteria, obtain informed consent, withdraw the blood samples, and record and manage the data.

Patients will be recruited before surgery. At the time the patient agrees to participate in the study, the functioning and adequate use of an intravenous patient-controlled analgesia (IV-PCA) pump will be explained by one of the members of the research team. The anesthetic, surgical, or postoperative care will not be affected by this research study.

Once the patient is in the theatre, standard intraoperative monitoring will be applied, including pulse oximetry, electrocardiography, automatic blood pressure cuff, capnography, and bispectral index monitoring (BIS system). The induction of anesthesia will be performed by the administration of remifentanil in a target-controlled infusion (TCI) using the MINTO model, propofol 1-2mg/kg and atracurium 0.5mg/kg or rocuronium 0.6mg/kg.

After induction, a second intravenous line will be installed in the contralateral arm exclusively to obtain blood samples. Subsequently, based on the ideal body weight, patients will receive a bolus of 0.1mg/kg of methadone at the beginning of surgery with a maximum dose of 20mg.

The maintenance of general anesthesia will be through the administration of sevoflurane to achieve BIS values between 40-60. Atracurium or rocuronium in doses of 5-10mg will be administered according to the neuromuscular block monitor and the infusion of remifentanil will be at the discretion of the anesthesiologist in charge to achieve mean arterial pressure within 20% of the baseline measure (previous induction of anesthesia). Episodes of hypotension will be treated with phenylephrine 50-100 mcg, ephedrine 6-12mg, or fluid bolus, as indicated.

Once the surgery is finished, the neuromuscular block will be reversed with neostigmine 30-70 mcg/kg or sugammadex 2-4mg/kg, as indicated and the patient will be extubated. Then, the patient will be transferred to the postoperative acute care unit (PACU) and assessed for pain by a nurse at the admission and every 15 minutes thereafter. If the patient reports a pain intensity greater than 3/10 at rest as measured by the numeric rating scale (NRS, being 0, no pain; 10, worst pain imaginable), methadone boluses of 3 mg will be administered every 15 minutes until the pain intensity is less than or equal to 3/10 or the patient has a respiratory rate less than 10/minute. Then, the IV-PCA device will be installed and its correct use will be explained again. The following IV-PCA program will be used: no background infusion, boluses of 1 milligram, and 8-minute lockout interval. Once the patient meets the discharge criteria from PACU using the Aldrete Scoring System (greater than or equal to 8 out of 10), the patient will be transferred to the ward.

In addition to the use of an IV-PCA device, the multimodal postoperative analgesia will consist of intravenous or oral paracetamol of 1gr every 8 hours as tolerated, rescue methadone boluses of 3 mg administered by the nurse in case the patient experiences pain intensity at rest greater than 3/10 despite an adequate use of the PCA pump. Also, no patient will receive non-steroidal anti-inflammatory drugs due to possible greater impairment of the baseline renal function. The pain team will remove the IV-PCA pump after 48 hours from the initial methadone bolus unless the surgical team determines earlier removal of the pump since the patient meets the discharge criteria from the hospital.

Number of blood samples: After the administration of methadone, a total of 12 venous blood samples will be obtained for each patient to investigate the potential accumulation of this opioid in the postoperative period. The samples will be collected at 5, 15, 30 and 60 minutes and 2, 4, 6, 9, 12, 24, 36, and/or 72 hours after the intraoperative bolus of methadone. The blood sample at 72 hours will be conditioned to the early removal of the IV-PCA pump in case the patient is ready to be discharged from the hospital. Blood samples will be collected in heparin tubes and centrifuged. The extracted serum will be placed in cryotubes which will be stored at -80°C until analysis. Methadone samples will be analyzed using a high-performance liquid chromatography (HPLC) spectrofluorometric method in the environmental and food analytical chemistry laboratory, Faculty of Chemistry and Pharmacy, Pontificia Universidad Católica de Chile. The lower limits of quantification (LLOQ) will be determined. Samples below the LLOQ will not be included in the analysis.

At the time of subsequent methadone plasma measurements, the following data will be recorded: IV-PCA boluses administered and demanded, pain intensity using the numeric rating scale, the degree of sedation using a 5-point scale, presence of pruritus/nausea/vomiting will also be recorded, and episodes of respiratory depression (respiratory rate <8/min) or oxygen saturation <90% measured by the pulse oximetry.

The nursing chart will also be reviewed to evaluate the additional administration of intravenous methadone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease (CrCl 15-60 ml/min)
* Patients over 18 years old undergoing surgery requiring general anesthesia with subsequent use of intravenous methadone patient-controlled analgesia
* Hospital stay ≥ 48 hours
* Body mass index 18-35 kg/m2

Exclusion Criteria:

* History of liver disease
* Need for dialysis (hemo or peritoneal dialysis)
* Use of home oxygen therapy
* American Society of Anesthesiologists (ASA) physical status IV-V
* Pregnancy
* Chronic opioid use
* Methadone allergy
* Prolonged QT interval
* Use of antiarrhythmics that prolong the QT interval
* Inability to understand the proper use of PCA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with a diagnosis of chronic kidney disease undergoing surgery requiring general anesthesia whose hospital stay is a minimum of 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration | 5, 15, 30, 60 minutes and 2, 4, 6, 9, 12, 24, 36 and 72 hours after the intraoperative bolus of methadone
  Blood samples will be taken, collected in heparin tubes, and centrifuged. The extracted serum will be placed in cryotubes that will be stored at -80 °C until analysis.
  Methadone samples will be analyzed using a high performance liquid chromatography (HPLC) spectrofluorometric method.
  Lower limits of quantification (LLOQ) will be determined and samples below the LLOQ will not be included in the analysis.

SECONDARY OUTCOMES:
Total use of methadone | 2, 4, 6, 9, 12, 24, 36 and 48 hours after the intraoperative bolus of methadone
  The administered and demanded boluses of the IV-PCA device will be assessed along with the intravenous methadone administered by the nursing staff.
Post-operative Pain | 2, 4, 6, 9, 12, 24, 36 and 48 hours after the intraoperative bolus of methadone
  The numeric rating scale will be used, being 0, no pain and 10, worst pain imaginable.
  If pain intensity is greater than 3 at rest, 3mg methadone boluses will be administered until an intensity of less than 3 is achieved or the patient presents a respiratory rate of less than 10/minute.
Nausea or vomiting | 2, 4, 6, 9, 12, 24, 36 and 48 hours after the intraoperative bolus of methadone
  Presence of nausea or vomiting in the postoperative acute care unit and the surgical ward.
Respiratory depression | 2, 4, 6, 9, 12, 24, 36 and 48 hours after the intraoperative bolus of methadone
  Presence of respiratory depression in the postoperative acute care unit and the surgical ward. The patient's clinical record will be reviewed.
  It will be considered as episodes of respiratory depression when the respiratory rate is less than 8/minute
Hypoxemia | 2, 4, 6, 9, 12, 24, 36 and 48 hours after the intraoperative bolus of methadone
  Presence of peripheral oxygen saturation less than 90%. The patient's clinical record will be reviewed.
Sedation | 2, 4, 6, 9, 12, 24, 36 and 48 hours after the intraoperative bolus of methadone
  The degree of sedation will be assessed using a five point sedation scale Score 1 (Barely arousable)= Asleep, needs shaking or shouting to arise Score 2 (Asleep)= Eyes closed, arousable with soft voice or light touch Score 3 (Sleepy)= Eyes opened, less active, and responsive Score 4= Awake Score 5= Agitated

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Vega, MD, Study Director — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Chile

REFERENCES:
- [Background] Kreek MJ, Schecter AJ, Gutjahr CL, Hecht M. Methadone use in patients with chronic renal disease. Drug Alcohol Depend. 1980 Mar;5(3):197-205. doi: 10.1016/0376-8716(80)90180-5. PMID 6986247
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Pharmacodynamics and pharmacokinetics of methadone during the perioperative period. Anesthesiology. 1982 Dec;57(6):458-67. doi: 10.1097/00000542-198212000-00005. No abstract available. PMID 6128949
- [Background] Inturrisi CE, Colburn WA, Kaiko RF, Houde RW, Foley KM. Pharmacokinetics and pharmacodynamics of methadone in patients with chronic pain. Clin Pharmacol Ther. 1987 Apr;41(4):392-401. doi: 10.1038/clpt.1987.47. PMID 3829576
- [Background] Sharma A, Tallchief D, Blood J, Kim T, London A, Kharasch ED. Perioperative pharmacokinetics of methadone in adolescents. Anesthesiology. 2011 Dec;115(6):1153-61. doi: 10.1097/ALN.0b013e318238fec5. PMID 22037641
- [Background] Davies G, Kingswood C, Street M. Pharmacokinetics of opioids in renal dysfunction. Clin Pharmacokinet. 1996 Dec;31(6):410-22. doi: 10.2165/00003088-199631060-00002. PMID 8968655
- [Background] Stemland CJ, Witte J, Colquhoun DA, Durieux ME, Langman LJ, Balireddy R, Thammishetti S, Abel MF, Anderson BJ. The pharmacokinetics of methadone in adolescents undergoing posterior spinal fusion. Paediatr Anaesth. 2013 Jan;23(1):51-7. doi: 10.1111/pan.12021. Epub 2012 Sep 14. PMID 22978825
- [Background] Yin OQ, Merante D, Truitt K, Miller R. Population pharmacokinetic modeling and simulation for assessing renal impairment effect on the pharmacokinetics of mirogabalin. J Clin Pharmacol. 2016 Feb;56(2):203-12. doi: 10.1002/jcph.584. Epub 2015 Sep 2. PMID 26138993
- [Background] Ji XW, Ji SM, He XR, Zhu X, Chen R, Lu W. Influences of renal function descriptors on population pharmacokinetic modeling of vancomycin in Chinese adult patients. Acta Pharmacol Sin. 2018 Feb;39(2):286-293. doi: 10.1038/aps.2017.57. Epub 2017 Aug 24. PMID 28836582
- [Background] Murphy GS, Szokol JW. Intraoperative Methadone in Surgical Patients: A Review of Clinical Investigations. Anesthesiology. 2019 Sep;131(3):678-692. doi: 10.1097/ALN.0000000000002755. No abstract available. PMID 31094758
- [Background] Kreutzwiser D, Tawfic QA. Methadone for Pain Management: A Pharmacotherapeutic Review. CNS Drugs. 2020 Aug;34(8):827-839. doi: 10.1007/s40263-020-00743-3. PMID 32564328